CLINICAL TRIAL: NCT01144858
Title: Clinical Value of Left Atrial Appendage Flow for Prediction of Successful Catheter Ablation for Persistent Atrial Fibrillation
Acronym: CLAAAF
Status: Terminated | Type: Observational
Why Stopped: 40 patients
Sponsor: Clinique Pasteur (Other)
Other Study IDs: past-1001-ryth
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2008-10

CONDITIONS: Persistent Atrial Fibrillation; Catheter Ablation
Keywords: atrial fibrillation; ablation catheter; left atrial appendage peak emptying velocity; tool for predicting successful catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with persistent atrial fibrillation ablation
  Interventions: Other: a complete transesophageal echocardiography

INTERVENTIONS:
Other: a complete transesophageal echocardiography — All patients were evaluated by a complete transesophageal echocardiography with multiplane probes with a 7-MHz transducer before catheter ablation .LA appendage flow was obtained by placing the pulsed Doppler sample volume at the orifice of the LA appendage, after which peak flow velocities were measured and averaged within each RR interval of 10 consecutive cardiac cycles

SUMMARY:
The purpose of this study was to determine whether left atrial appendage flow velocity, as determined using trans esophageal echocardiography (TEE), predicts the outcome after catheter ablation of persistent Atrial fibrillation( pAF).

DETAILED DESCRIPTION:
40 PAF patients underwent 3D mapping and ablation. A stepwise approach including circumferential pulmonary vein (PV) isolation, continuous complex-fractionated electrogram (CFE) ablation and linear ablation was performed by the same operator. The procedural end point was termination of persistent AF by catheter ablation, either by conversion directly to sinus rhythm or to atrial tachycardia. Left atrial appendage (LAA) peak flow velocities were measured with transesophageal echography and averaged within each RR interval of 10 consecutive cardiac cycles.

ELIGIBILITY:
Inclusion Criteria:

* First-time radiofrequency catheter ablation for pAF. pAF was defined as continuous AF lasting longer than 1 month, resistant to either electrical or pharmacological cardioversion.
* Informed consent

Exclusion Criteria:

* Severe valvular disease requiring surgery
* Valvular prosthesis
* Known severe coronary artery disease
* Atrial and/or ventricular thrombosis
* New York Heart Association functional class III to IV
* Cerebrovascular disease
* Pulmonary embolism
* Latent or manifest hyperthyroidism

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 40 consecutive patients who underwent first-time radiofrequency catheter ablation for pAF. pAF was defined as continuous AF lasting longer than 1 month, resistant to either electrical or pharmacological cardioversion
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-01; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
termination of persistent AF by catheter ablation

SECONDARY OUTCOMES:
Recurrences of AF were therefore determined from holter monitoring at 3 and 6 months or 12 leads ECG in care of symptomatic palpitation with clinical interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Pasteur, Toulouse, 43-45 Avenue de Lombez, France

REFERENCES:
- [Derived] Combes S, Jacob S, Combes N, Karam N, Chaumeil A, Guy-Moyat B, Treguer F, Deplagne A, Boveda S, Marijon E, Albenque JP. Predicting favourable outcomes in the setting of radiofrequency catheter ablation of long-standing persistent atrial fibrillation: a pilot study assessing the value of left atrial appendage peak flow velocity. Arch Cardiovasc Dis. 2013 Jan;106(1):36-43. doi: 10.1016/j.acvd.2012.09.002. Epub 2012 Dec 20. PMID 23374970